CLINICAL TRIAL: NCT02758717
Title: Phase II, Multi-Center Trial of Nivolumab and Brentuximab Vedotin in Patients With Untreated Hodgkin Lymphoma Over the Age of 60 Years or Unable to Receive Standard Adriamycin, Bleomycin, Vinblastine, and Dacarbazine (ABVD) Chemotherapy
Brief Title: Nivolumab and Brentuximab Vedotin in Treating Older Patients With Untreated Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RU051505I; NCI-2016-00468 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RU051505I (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2016-04-12; First posted 2016-05-02 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Ann Arbor Stage IB Hodgkin Lymphoma; Ann Arbor Stage II Hodgkin Lymphoma; Ann Arbor Stage IIA Hodgkin Lymphoma; Ann Arbor Stage IIB Hodgkin Lymphoma; Ann Arbor Stage III Hodgkin Lymphoma; Ann Arbor Stage IIIA Hodgkin Lymphoma; Ann Arbor Stage IIIB Hodgkin Lymphoma; Ann Arbor Stage IV Hodgkin Lymphoma; Ann Arbor Stage IVA Hodgkin Lymphoma; Ann Arbor Stage IVB Hodgkin Lymphoma; Classic Hodgkin Lymphoma
MeSH Terms: interventions — Brentuximab Vedotin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (brentuximab vedotin, nivolumab) (Experimental): Patients receive brentuximab vedotin IV over 30 minutes and nivolumab IV over 60 minutes on day 1. Treatment repeats every 21 days for 7 cycles and 6-8 weeks in cycle 8 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Biological: Nivolumab

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies how well nivolumab and brentuximab vedotin work in treating older patients with untreated Hodgkin lymphoma. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Biological therapies, such as brentuximab vedotin, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Nivolumab and brentuximab vedotin may work better in treating older patients with untreated Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy based on overall metabolic response rate (partial metabolic response [PMR] + complete metabolic remission [CMR]) of brentuximab vedotin/nivolumab in previously untreated Hodgkin lymphoma patients 60 years of age or older, or those considered unsuitable for standard chemotherapy because of a low cardiac ejection fraction (< 50%) or impaired pulmonary or renal function.

SECONDARY OBJECTIVES:

I. The complete metabolic response (CMR) rate. II. Safety and tolerability of the regimen in this patient population. III. Duration of response (DOR). IV. Progression-free survival (PFS). V. Overall survival (OS).

CORRELATIVE RESEARCH OBJECTIVES:

I. T-cell/cytokine - peripheral blood specimens will be used to assess T-cell activation and cytokine up regulation as measures of treatment effect.

II. Biomarkers - intratumoral cell populations, genetic variability, serum cytokines and T-cell activation will be evaluated to identify potential biomarkers that correlate with response to therapy.

OUTLINE:

Patients receive brentuximab vedotin intravenously (IV) over 30 minutes and nivolumab IV over 60 minutes on day 1. Treatment repeats every 21 days for 7 cycles and 6-8 weeks in cycle 8 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 30 days for 90 days, every 90 days for 2.5 years, and then every 6 months until 5 years from registration.

ELIGIBILITY:
Inclusion Criteria:

* Classical Hodgkin lymphoma determined by local hematopathology review
* One of the following:

  * Age >= 60 years
  * Age < 60 years but unsuitable for standard chemotherapy because of a cardiac ejection fraction of < 50%, a pulmonary diffusion capacity < 80%, or a creatinine clearance >= 30 and < 60 mL/min, or refused standard chemotherapy despite efforts to convince them otherwise
* Requirement for systemic chemotherapy: all stages except IA (not bulky disease), if involved field is considered radiotherapy (RT) curative
* Previously untreated with either chemotherapy, radiation therapy or either brentuximab vedotin or nivolumab, or another check point inhibitor
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1500/mm^3, unless secondary to bone marrow involvement; obtained =< 7 days prior to registration
* Leukocytes >= 3,000/mm^3, obtained =< 7 days prior to registration
* Platelet count >= 100,000/mm^3, obtained =< 7 days prior to registration
* Hemoglobin > 9.0 g/dL - unless determined by treating physician to be disease related, obtained =< 7 days prior to registration
* Total bilirubin =< 1.5 x upper limit of normal (ULN), obtained =< 7 days prior to registration
* Aspartate aminotransferase (aspartate transaminase [AST]) =< 2.5 x ULN, obtained =< 7 days prior to registration
* Alanine aminotransferase (alanine transaminase [ALT]) =< 2.5 x ULN, obtained =< 7 days prior to registration
* Creatinine =< 2.0 mg/dL, obtained =< 7 days prior to registration
* Amylase and/or lipase =< 1.5 x ULN, obtained =< 7 days prior to registration
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to registration

  * Note: women of child-bearing potential (WOCBP) must use appropriate method(s) of contraception; WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug; men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year; men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product; women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

  * Note: during the active monitoring phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Ability to understand and willingness to sign an informed written consent
* Provide blood and tissue samples for mandatory correlative research purposes

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Active, known or suspected autoimmune disease; note: subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Use of systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications =< 14 days of registration; Note: Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Immunocompromised patients, patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) and currently receiving antiretroviral therapy, patients with a prior history of known or suspected autoimmune disease, active hepatitis B virus surface antigen (HBV sAg+), active hepatitis C (if antibody [Ab]+ then polymerase chain reaction [PCR]+) indicating acute or chronic infection, and/or history of interstitial lung disease
* Allergy to brentuximab vedotin and/or nivolumab
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Have had prior chemotherapy or radiotherapy for Hodgkin lymphoma
* Have received either of the study drugs
* < 60 years who are considered candidates for standard chemotherapy
* >= grade 2 peripheral neuropathy
* Other active malignancy =< 2 years prior to registration, unless treated with curative intent; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer
* Active central nervous system (CNS) involvement or leptomeningeal metastases involvement
* Known history of pancreatitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2025-09-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Cheson, Principal Investigator — Academic and Community Cancer Research United
Locations (9):
- United States (9):
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Cheson BD, Bartlett NL, LaPlant B, Lee HJ, Advani RJ, Christian B, Diefenbach CS, Feldman TA, Ansell SM. Brentuximab vedotin plus nivolumab as first-line therapy in older or chemotherapy-ineligible patients with Hodgkin lymphoma (ACCRU): a multicentre, single-arm, phase 2 trial. Lancet Haematol. 2020 Nov;7(11):e808-e815. doi: 10.1016/S2352-3026(20)30275-1. Epub 2020 Oct 1. PMID 33010817

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Brentuximab Vedotin, Nivolumab): Patients receive 1.8 mg/kg (cap at 180 mg) in 100 to 250 mL NS to final concentration 0.4 mg/mL to 1.8 mg/mL brentuximab vedotin IV over 30 minutes and 3 mg/kg in 100 cc NS nivolumab IV over 60 minutes on day 1. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Brentuximab Vedotin, Nivolumab)
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Brentuximab Vedotin, Nivolumab)
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 71.5 [46.0 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 39
  More than one race | 0
  Unknown or Not Reported | 3
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 14
    1 | 26
    2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Metabolic Response Rate
Description: The primary endpoint of this trial is the rate (percentage) of overall metabolic response. A metabolic response is defined as a participant who has achieved an objective status of Partial metabolic response (PMR) or Complete metabolic response (CMR) at the end of cycle 8. Response is based on PET/CT based on the revised 2014 Lugano Classification. (PMR: Score 4 (uptake moderately > liver) or 5 (uptake markedly higher than liver and/or new lesions) with reduced uptake compared with baseline and residual mass(es) of any size CMR: Score 1 (no uptake above background), 2 (uptake<=mediastinum), or 3 (uptake > mediastinum but <= liver) with or without a residual mass on PET Deauville 5-Point-Scale. The scale ranges from 1 to 5, where 1 is best and 5 is the worst.
Time Frame: Up to 8 cycles of treatment (approximately 29 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Brentuximab Vedotin, Nivolumab)
Number analyzed (Participants) | 46
percentage of participants | 60.9 [45.4 to 74.9]

2. Secondary Outcome: Number of Participants With an Overall Response of Complete Metabolic Response
Description: The number of participants with an overall response of Complete metabolic response. Response is based on PET/CT based on the revised 2014 Lugano Classification. (CMR: Score 1 (no uptake above background), 2 (uptake<=mediastinum), or 3 (uptake > mediastinum but <= liver) with or without a residual mass on PET Deauville 5-Point-Scale. The scale ranges from 1 to 5, where 1 is best and 5 is the worst.
Time Frame: Up to end of course 8
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Brentuximab Vedotin, Nivolumab)
Number analyzed (Participants) | 46
Participants | 22

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR is time from the date at which the patient's objective status is first noted to be a CMR or PMR to the earliest date progression (progressive metabolic disease [PMD] or progressive disease [PD]) is documented. Response is based on PET/CT based on the revised 2014 Lugano Classification. (PMR: Score 4 (uptake moderately > liver) or 5 (uptake markedly higher than liver and/or new lesions) CMR: Score 1 (no uptake above background), 2 (uptake<=mediastinum), or 3 (uptake > mediastinum but <= liver) with or without a residual mass on PET Deauville 5-Point-Scale. The scale ranges from 1 to 5, where 1 is best and 5 is the worst. PMD: Score 4 or 5 with an increase in intensity of uptake from baseline and/or New FDG-avid foci consistent with lymphoma at interim or end-of-treatment assessment PD: An individual node/lesion must be abnormal with: LDi > 1.5 cm and Increase by ≥ 50% from PPD nadir and, An increase in LDi or SDi from nadir, 0.5 cm for lesions ≤2 cm, 1.0 cm for lesions > 2 cm)
Time Frame: 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Brentuximab Vedotin, Nivolumab)
Number analyzed (Participants) | 46
months | NA [11.1 to NA] — Median and upper limit duration of response were not estimatable due to a lack of events. Insufficient number of participants with events

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from registration to the earliest date of documentation of disease progression (Progressive metabolic disease (PMD) or Progressive disease (PD)) or death due to any cause. Response is based on PET/CT based on the revised 2014 Lugano Classification. (PMD: Score 4 or 5 with an increase in intensity of uptake from baseline and/or New FDG-avid foci consistent with lymphoma at interim or end-of-treatment assessment PD: An individual node/lesion must be abnormal with: LDi > 1.5 cm and Increase by ≥ 50% from PPD nadir and, An increase in LDi or SDi from nadir, 0.5 cm for lesions ≤2 cm, 1.0 cm for lesions > 2 cm)
Time Frame: 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Brentuximab Vedotin, Nivolumab)
Number analyzed (Participants) | 46
months | 18.3 [12.7 to NA] — The upper limit of the confidence interval was not reached due to a lack of events. Insufficient number of participants with events.

5. Secondary Outcome: Overall Survival
Description: The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Time Frame: 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Brentuximab Vedotin, Nivolumab)
Number analyzed (Participants) | 46
months | NA [NA to NA] — Median overall survival time was not estimatable due to the low number of patient deaths

6. Secondary Outcome: Number of Participants Experiencing at Least One Adverse Events Graded 3 or Higher Deemed at Least Possibly Related to Treatment
Description: Number of participants experiencing at least one toxicity. Toxicity is defined as an adverse event graded 3 or higher by Common Terminology Criteria for Adverse Events version 4.0 deemed at least possibly related to treatment.
Time Frame: Up to 8 cycles of treatment (approximately 29 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Brentuximab Vedotin, Nivolumab)
Number analyzed (Participants) | 46
Participants | 30

ADVERSE EVENTS:
Time Frame: 30 months
Arm/Group | Treatment (Brentuximab Vedotin, Nivolumab)
All-Cause Mortality (participants affected / at risk) | 4/46
Serious Adverse Events (participants affected / at risk) | 21/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Brentuximab Vedotin, Nivolumab) (N=46)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 4 (4)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Serum amylase increased (Investigations) | 2 (2)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Brentuximab Vedotin, Nivolumab) (N=46)
Anemia (Blood and lymphatic system disorders) | 4 (6)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (9)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (8)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (4)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (5)
Nausea (Gastrointestinal disorders) | 8 (10)
Rectal fistula (Gastrointestinal disorders) | 1 (2)
Fatigue (General disorders) | 15 (34)
Fever (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 3 (4)
Papulopustular rash (Infections and infestations) | 1 (3)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (6)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (8)
Alanine aminotransferase increased (Investigations) | 4 (9)
Aspartate aminotransferase increased (Investigations) | 3 (8)
Creatinine increased (Investigations) | 12 (35)
Ejection fraction decreased (Investigations) | 1 (1)
GGT increased (Investigations) | 1 (1)
INR increased (Investigations) | 2 (4)
Investigations - Other, specify (Investigations) | 1 (1)
Lipase increased (Investigations) | 6 (16)
Lymphocyte count decreased (Investigations) | 5 (24)
Neutrophil count decreased (Investigations) | 19 (57)
Platelet count decreased (Investigations) | 15 (61)
Serum amylase increased (Investigations) | 6 (10)
Weight gain (Investigations) | 1 (2)
Weight loss (Investigations) | 2 (8)
White blood cell decreased (Investigations) | 24 (76)
Anorexia (Metabolism and nutrition disorders) | 2 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (8)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (22)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (6)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 17 (96)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (40)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 (62)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (17)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (19)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 10 (33)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT02758717/Prot_SAP_000.pdf